CLINICAL TRIAL: NCT05426616
Title: A Randomized Controlled Trial Comparing Titanium Reinforced d-PTFE Membrane to Collagen Membrane for Guided Bone Regeneration at Single Tooth Sites in the Premaxilla: a Clinical, CBCT and Histomorphometric Analysis
Brief Title: Titanium Reinforced d-PTFE Membrane Versus Collagen Membrane For Guided Bone Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-11825
Record Dates: First submitted 2022-06-11; First posted 2022-06-22 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Ridge Enlargement
Keywords: Guided bone regeneration; Resorbable collagen membrane; Titanium reinforced d-PTFE membrane

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Collagen membrane (Active Comparator): (Xenoprotect, Nobel Biocare, Göteborg, Sweden)
  Interventions: Device: collagen membrane (Creos Xenoprotect , Nobel Biocare AB, Göteborg, Sweden)
- Test group: titanium reinforced d-PTFE membrane (Experimental): (Creos Syntoprotect,Nobel Biocare AB, Göteborg, Sweden)
  Interventions: Device: titanium reinforced d-PTFE membrane (Creos Syntoprotect , Nobel Biocare AB, Göteborg, Sweden)

INTERVENTIONS:
Device: collagen membrane (Creos Xenoprotect , Nobel Biocare AB, Göteborg, Sweden) — A mucoperiosteal flap will be raised with two vertical releasing on each side of the edentulous space. Autogenous bone chips are harvested from the retromolar area with bone scrapers and/or from an edentulous site using ACM bone collector. DBBM particles soaked in blood are mixed with autogenous bone chips to a ratio of 1:1. After having made multiple bone perforations at the buccal aspect of the recipient site, the mixture of bone chips and DBBM is applied. An individualized collagen membrane is attached on top using membrane fixation pins. Prior to fixation of the final pin, bone grafting material is additionally applied from the lateral aspect to ensure that it is properly packed under the membrane and fully stable. Following release of the periosteum and muscle insertion, tension-free primary wound closure is achieved.
  Arms: Control group: Collagen membrane
Device: titanium reinforced d-PTFE membrane (Creos Syntoprotect , Nobel Biocare AB, Göteborg, Sweden) — A mucoperiosteal flap will be raised with two vertical releasing on each side of the edentulous space. Autogenous bone chips are harvested from the retromolar area with bone scrapers and/or from an edentulous site using ACM bone collector. DBBM particles soaked in blood are mixed with autogenous bone chips to a ratio of 1:1. After multiple bone perforations at the buccal aspect of the recipient site, the mixture of bone chips and DBBM is applied.A titanium reinforced d-PTFE membrane is attached on top using membrane fixation pins. Care is taken to leave a distance of at least 1 mm between the membrane and neighboring teeth. Prior to fixation of the final pin, bone grafting material is additionally applied from the lateral aspect to ensure that it is properly packed under the membrane and fully stable. Following release of the periosteum and muscle insertion, tension-free primary wound closure is achieved. The membrane is removed after 9 months, prior to implant placement.
  Arms: Test group: titanium reinforced d-PTFE membrane

SUMMARY:
After tooth extraction, shrinkage of the bone is expected with 50% reduction of alveolar width. Patients at least 3months after tooth extraction and in need of single oral implant placement in the anterior maxilla with both neighboring teeth present, were invited to participate in an inter-subject RCT if insufficient residual alveolar bone was left for proper implant placement. Guided bone regeneration has been used to recreate bone volume. A combination of xenogenous bone (Creos Xenogain , Nobel Biocare AB, Göteborg, Sweden) and autologous bone chips in a 1:1 ratio, is protected by a membrane fixated in the bone. A resorbable, non-stable membrane (Creos Xenoprotect, Nobel Biocare AB, Göteborg, Sweden) or non-resorbable titanium reinforced d-PTFE membrane (Creos Syntoprotect , Nobel Biocare AB, Göteborg, Sweden) can be used.

This study aims to compare the effectivity of the two membranes by measuring changes in bone dimensions. The resorbable membrane has the advantage that it does not need to be removed, whereas the titanium reinforced membrane can protect the rebuilt volume better against external forces.

Patients start to take systemic antibiotics (Amoxicilline 1g) and anti-inflammatory medication (ibuprofen 600 mg) 1h pre-operatively. Following local anesthesia (Septanest special, Septodont, Saint Maur des Fossés, France) and oral disinfection (Corsodyl mouth rinse, GSK, Wavre, Belgium), a large mucoperiosteal flap will be raised with two vertical releasing on each side of the edentulous space and at the distal aspect of the second neighboring tooth. The flap extends to the base of the alveolar process to allow full access. Autogenous bone chips are harvested from the retromolar area with bone scrapers and/or from an edentulous site using ACM bone collector (NeoBiotech, Guro-gu Seoul, Republic of Korea). DBBM particles (Xenogain, Nobel Biocare, Göteborg, Sweden) soaked in blood are mixed with autogenous bone chips to a ratio of 1/1. After having made multiple bone perforations at the buccal aspect of the recipient site, the mixture of bone chips and DBBM is applied. An individualized collagen membrane (Xenoprotect, Nobel Biocare, Göteborg, Sweden) or a non-resorbable titanium reinforced d-PTFE membrane is attached on top using membrane fixation pins. Prior to fixation of the final pin, bone grafting material is additionally applied from the lateral aspect to ensure that it is properly packed under the membrane and fully stable. Following release of the periosteum and muscle insertion, tension-free primary wound closure is achieved with horizontal mattress 4/0 titanium reinforced d-PTFE sutures and single 6/0 monofilament sutures. Patients continue the intake of antibiotics and anti-inflammatory medication for 7 days and use an oral mouthrinse during 2 weeks. Sutures are removed after 2 weeks, and an implant is installed after 9 months following 3D implant planning.

A sample size calculation indicated 17 patients to be included per group. To compensate for one drop-out, 18 patients would be treated with collagen membrane and 18 would be treated with titanium reinforced d-PTFE.

Changes in horizontal bone dimensions over time is the primary outcome. Prior to surgery, immediately after GBR, at 9 months, at 3 years and 5 years a CBCT is taken. Every CBCT is superimposed to the baseline CBCT in designated software and horizontal buccal bone dimensions are measured.

Secondary outcomes include

* Membrane exposure
* Intrasurgical changes in bone crest width over time
* Intrasurgical assessment of bone quality at implant placement at the palatal, midcrestal and buccal aspect
* Need for re-grafting at implant placement
* Need for soft tissue grafting at implant placement
* Need for augmentation of keratinized mucosa at implant placement
* Volumetric increase in buccal bone at 3 and 5 years
* Peri-implant health at 3 and 5 years by means of intra-oral radiograph
* Esthetic outcomes at 3 and 5 years
* Histomorphometric analysis on 20 cases (10 per group)

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene defined as full-mouth plaque score ≤ 25% (O'Leary et al. 1972)
* presence of a single tooth gap in the anterior maxilla (15-25) with both neighboring teeth present
* failing tooth at least 3 months earlier removed

Exclusion Criteria:

* systemic diseases
* smoking; (history of) periodontal disease
* untreated caries lesions
* pregnancy (will be explicitly asked)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in horizontal bone dimensions over time | baseline = t0, immediately after GBR = t1, at 9 months= t2, 3 years = t3 and 5 years=t4
  At T0, t1, t2, t3 and t4 a CBCT is taken. Every CBCT is superimposed to the baseline CBCT in designated software and horizontal buccal bone dimensions are measured at 1 mm, 3 mm, 5 mm, 7 mm and 9 mm from the crest. The changes from baseline in horizontal bone dimensions at the different levels is calculated.

SECONDARY OUTCOMES:
Membrane exposure | During the 9 months of healing after GBR.
  Wound dehiscence after GBR could expose the membrane. Clinically assessment if the membrane is coming exposed through the mucosa during the healing period of 9months after placement, results in a % of cases with membrane exposure.
Intrasurgical changes in bone crest width over time | Baseline, after GBR and 9 months after GBR during implant placement procedure.
  Measurement of the bone crest width intrasurgically, after mucoperiosteal flap preparation.
Bone type: clinician perception (hand feel resistance) | t2 = 9 months after GBR, at implant placement
  Classification by Misch. Tactile sense of the surgeon in the assessment of bone density, groups (D1-D4). D1 bone type = homogenous dense cortical. D2 = combination of dense-to-porous cortical bone on the crest and trabecular bone from 40% to 60% on the inside. D3 = thinner porous cortical bone on the crest and fine trabecular bone within the ridge. D4 = bone has the least trabecular density with little or no cortical crestal bone.
Bone dimensions vertically and horizontally | t2 = 9 months after GBR, at implant placement
  Bone volume assessment for the ideal restorative driven position of the implant after 9 months of healing, reporting if insufficient bone was leading to additional bone grafting simultaneously at the time of implant placement.
  Edentulous bone ridge classification followed three-dimensional (3D) quantity of alveolar bone shape and volume based on CBCT measurements. (UCLA) Classification: Type I: sufficient alveolar shape for implants, Type II: insufficient alveolar bone on the buccal site, Type III: knife edge shape with sufficient alveolar bone height, Type IV: insufficient alveolar bone height.
Buccal soft tissue thickness | t2 = 9 months after GBR, at implant placement
  Buccal concavity after resorption of the soft tissue, can cause additional need for soft tissue augmentation procedure. The need for soft tissue augmentation will be scored by the clinician. The thickness of the soft tissues was measured (in mm) at t2 (9months after GBR), t3 (3 years) and T4 (5years) perpendicular to the long axis of the implant. Buccal soft tissue thickness was measured from the bone-soft tissue interface to the buccal soft tissue outline at the same levels as horizontal bone dimensions.
Buccal keratinized soft tissue width | t2 = 9 months after GBR, at implant placement
  The width of the keratinized soft tissues buccally was measured clinically (in mm) at t2 (9months after GBR), t3 (3 years) and T4 (5years) from the gingival margin to mucogingival junction. Minimally 3 mm provides a prosthetic friendly environment, allows oral hygiene maintenance, resists recession, and enhances esthetic blending. If less than 3mm, additional soft tissue grafting can be indicated.
Volumetric changes in buccal bone at 3 and 5 years | baseline = t0, immediately after GBR = t1, at 9 months= t2, 3 years = t3 and 5 years=t4
  Volumetric measurement with CBCT by superimposed the images in specialized software (OnDemand3D, Cybermed Inc., Seoul, South-Korea). Changes in bone volume are calculated by subtracting.
Peri-implant health | At 3 and 5 years
  Evaluation by means of intra-oral radiograph of bone level.
Pink Esthetic Score | At 3 and 5 years
  The PES awards 7 parameters: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue colour, soft tissue texture. Each parameter is assessed with a 0-1-2 score, yielding a PES score ranging from 0 (worst aesthetic outcome) to 14 (perfect aesthetic outcome).
Histomorphometric analysis | t2 = 9 months after GBR, at implant placement
  On 20 cases (10 per group), with a trepan bur, bone samples are removed and collected from implant site at 9 months right before implant placement, for measurements: Vital bone fraction, biomaterial fraction, connective tissue fraction and cell counts.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Cosyn, Professor, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Centrum voor Parodontologie en Orale Implantologie, Zottegem, Oost-Vlaanderen
  - Parodonto, Zwijnaarde, Oost-Vlaanderen

REFERENCES:
- [Derived] Hindryckx M, De Bruyckere T, Hitz-Steiger S, Seyssens L, Shtino R, Younes F, Thoma D, Cosyn J. A Multi-Center RCT Comparing Titanium-Reinforced dPTFE Membrane to Collagen Membrane in Horizontal Bone Augmentation at Single Sites in the Anterior Maxilla: Clinical and Histological Outcomes. Clin Implant Dent Relat Res. 2025 Dec;27(6):e70097. doi: 10.1111/cid.70097. PMID 41185408
- [Derived] Hindryckx M, De Bruyckere T, De Buyser S, Seyssens L, Shtino R, Younes F, Cosyn J. A Multi-Centre Randomised Controlled Trial Comparing dPTFE Membrane to Collagen Membrane in Lateral Bone Augmentation at Single Sites in the Anterior Maxilla: 1-Year Results. J Clin Periodontol. 2025 Aug;52(8):1136-1146. doi: 10.1111/jcpe.14174. Epub 2025 Apr 29. PMID 40298001